CLINICAL TRIAL: NCT01505153
Title: Phase I Trial of Intratumoral Bi-functional shRNA Stathmin 1-knockdown Lipoplex in Patients With Advanced and/or Metastatic Cancer
Brief Title: Phase I Intratumoral Pbi-shRNA STMN1 LP in Advanced and/or Metastatic Cancer
Acronym: STMN1-LP
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gradalis, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CL-PTL 103
Record Dates: First submitted 2012-01-04; First posted 2012-01-06 (Estimated); Last update posted 2018-02-22 (Actual); Status verified 2018-02

CONDITIONS: Advanced Cancer; Metastatic Cancer; Solid Tumors
Keywords: Advanced cancer; Metastatic cancer; solid tumors; Melanoma
MeSH Terms: conditions — Neoplasm Metastasis; Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- pbi-shRNA STMN1 LP (Experimental): pbi-shRNA™ STMN1 LP administered by a single intratumoral (IT) injection.
  Interventions: Biological: pbi-shRNA STMN1 LP

INTERVENTIONS:
Biological: pbi-shRNA STMN1 LP — This is a Phase I safety trial of bifunctional shRNA-STMN1 (pbi-shRNA™STMN1) BIV (bilamellar invaginated vesicle) lipoplex (LP), pbi-shRNA™ STMN1 LP administered by a single intratumoral (IT) injection. Patients will accrue in 4-patient escalation cohorts using a modified Fibronacci escalation schema at a starting intratumoral dose of 0.010 mg/kg of DNA through a dose of 0.053 mg/kg DNA intratumoral / single dose.

SUMMARY:
This is a Phase I safety trial of bifunctional shRNA-STMN1 (pbi-shRNA™STMN1) BIV (bilamellar invaginated vesicle) lipoplex (LP), pbi-shRNA™ STMN1 LP administered by a single intratumoral (IT) injection. Patients with superficially accessible advanced cancer following prior therapies will be entered into the study following a modified dose escalation design based on the demonstrated safety of our previous clinical experience (BB-IND 13744) with the same liposome and vector DNA backbone expressing a different transgene (of which doses up to 7 mg DNA IV/single dose have been administered). Patients will accrue in 4-patient escalation cohorts using a modified Fibronacci escalation schema (100%-50%-33%-33%) at a starting intratumoral dose of 0.010 mg/kg of DNA through a dose of 0.053 mg/kg DNA intratumoral / single dose. Should a single, but not more than two (2), ≥ Grade 3 Dose Limiting Toxicity (DLT) occur in any cohort, following mandated review (see below) an additional two (2) patients will be accrued at that dose (total of six). If more than one ≥ Grade 3 toxicity occurs in any cohort, the preceding dose cohort will be expanded to six (from four) and if < 2/6 patients experience ≥ Grade 3 toxicity, that dose will be the Phase II recommended dose. Should no ≥ Grade 3 toxicity occur in any cohort (other than Grade 3 local injection site reaction), an additional two (2) patients will be treated at 0.053 mg/kg DNA intratumoral / single dose.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed advanced and/or metastatic cancer, and, if limited to a single lesion, not considered a candidate for curative surgery or radiation therapy).
2. Biopsy accessible lesion.
3. Per cohort dose/volume, the volume of the lesion to be injected must be 3x volume of the injectate.
4. Subjects that have completed all acceptable therapies with curative potential that are the current standard of care for their respective diseases.
5. Recovered from all toxicities (≤ Grade 1) related to prior therapies except for alopecia.
6. 1 measurable or evaluable lesion; ≥ 1.8 cm diameter for cohort 1 (see Table 10); injection and biopsy accessible.
7. Age ≥18 years.
8. ECOG performance status (PS) 0-2.
9. Organ and marrow function as defined below:

   Absolute granulocyte count ≥ 1,500/mm^3 Platelets ≥ 100,000/mm^3 Total bilirubin ≤ 1.5x institutional ULN Creatinine ≤ 2.0 mg/dL
10. Ability to understand and the willingness to sign a written informed consent document including permission for pre- and Days 1 and 2 post- injection biopsy and Day 8 injected lesion excision.
11. Negative pregnancy test.

Exclusion Criteria:

1. Surgery involving general anesthesia, chemotherapy, radiotherapy, or immunotherapy within 3 weeks prior to entering the study.
2. Patient must not have received any other investigational agents within 4 weeks prior to study entry.
3. Patients with known brain metastases unless treated with whole brain radiation and stable for >/= 2 months or treated with stereotactic radiotherapy only and stable for >/=1 month.
4. Short term (<30 days) concurrent systemic steroids ≤0.125 mg/kg prednisone per day (maximum 7.5 mg/day) and bronchodilators (inhaled steroids) are permitted; other steroid regimens and/or immunosuppressives are excluded.
5. Prior malignancy (excluding nonmelanoma carcinomas of the skin) unless in remission for >/= 2 years.
6. Kaposi's Sarcoma.
7. Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
8. Patients who are pregnant or nursing.
9. Patients with known HIV.
10. Patients with chronic Hepatitis B and C infection.
11. Patients with uncontrolled diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-02 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-04-13 (Actual)

PRIMARY OUTCOMES:
To determine the safety of intratumoral administration of pbi-shRNA™ STMN1 LP | 1 month
  To determine the safety of intratumoral administration of pbi-shRNA™ STMN1 LP in patients with superficial advanced and/or metastatic cancer who have no acceptable form of standard therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Minal Barve, MD, Principal Investigator — Mary Crowley Cancer Research Centers
Locations (1):
- Mary Crowley Cancer Research Centers, Dallas, Texas, United States

REFERENCES:
- [Background] Phadke AP, Jay CM, Wang Z, Chen S, Liu S, Haddock C, Kumar P, Pappen BO, Rao DD, Templeton NS, Daniels EQ, Webb C, Monsma D, Scott S, Dylewski D, Frieboes HB, Brunicardi FC, Senzer N, Maples PB, Nemunaitis J, Tong AW. In vivo safety and antitumor efficacy of bifunctional small hairpin RNAs specific for the human Stathmin 1 oncoprotein. DNA Cell Biol. 2011 Sep;30(9):715-26. doi: 10.1089/dna.2011.1240. Epub 2011 May 25. PMID 21612405
- [Background] Rao DD, Maples PB, Senzer N, Kumar P, Wang Z, Pappen BO, Yu Y, Haddock C, Jay C, Phadke AP, Chen S, Kuhn J, Dylewski D, Scott S, Monsma D, Webb C, Tong A, Shanahan D, Nemunaitis J. Enhanced target gene knockdown by a bifunctional shRNA: a novel approach of RNA interference. Cancer Gene Ther. 2010 Nov;17(11):780-91. doi: 10.1038/cgt.2010.35. Epub 2010 Jul 2. PMID 20596090
- [Background] Rana S, Maples PB, Senzer N, Nemunaitis J. Stathmin 1: a novel therapeutic target for anticancer activity. Expert Rev Anticancer Ther. 2008 Sep;8(9):1461-70. doi: 10.1586/14737140.8.9.1461. PMID 18759697